CLINICAL TRIAL: NCT02679638
Title: Factors and Perceptions Affecting Treatment Choices of Breast Cancer Patients. Multi-center Cross-sectional Study in Israel Among Breast Cancer Survivors, With a Preliminary Qualitative Study
Brief Title: Factors and Perceptions Affecting Treatment Choices of Breast Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Haifa (Other)
Responsible Party: Sponsor
Other Study IDs: 27-15
Record Dates: First submitted 2016-02-04; First posted 2016-02-10 (Estimated); Last update posted 2016-02-10 (Estimated); Status verified 2016-02

CONDITIONS: Breast Cancer
Keywords: breast cancer; treatment choice; factor; perception
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Kaplan Hospital: Breast cancer survivors recruited at the Kaplan Medical Center
  Interventions: Other: Factors and perceptions questionnaire; Other: Qualitative interview
- Rambam Hospital: Breast cancer survivors recruited at the Rambam Medical Center
  Interventions: Other: Factors and perceptions questionnaire; Other: Qualitative interview
- Sheba: Breast cancer survivors recruited at the Sheba Medical Center
  Interventions: Other: Factors and perceptions questionnaire
- Barzilai: Breast cancer survivors recruited at the Barzilai Medical Center
  Interventions: Other: Factors and perceptions questionnaire

INTERVENTIONS:
Other: Factors and perceptions questionnaire — A detailed questionnaire inquiring about demand factors, supply factors and perceptions affecting patients' treatment choices in 5 key decision points: participation role in the decision making process, hospital choice, treatment regimen choice, surgical extent and surgeon choice.
Other: Qualitative interview — Depth interviews with 20 breast cancer patients, 2 spouses and 3 staff members.
  Groups: Kaplan Hospital; Rambam Hospital

SUMMARY:
A Multi-center Cross-sectional quantitative study with a preliminary qualitative study part aiming to identify and analyze demand factors, supply factors and perceptions affecting Breast Cancer patients' treatment choices of Breast Cancer patients in 5 key decision points: participation role in the decision making process, hospital choice, treatment regimen choice, surgical extent and surgeon choice. 25 patients and caregivers will participate in the qualitative part and 425 Israeli Breast Cancer patients will participate in the quantitative study.

DETAILED DESCRIPTION:
Background:

Breast Cancer (BC) is the most common cancer in women worldwide. Newly diagnosed BC patients are asked to participate in a number of treatment related decisions. No research has systematically studied the full decision sequence in a disease such as BC, analyzing demand factors, supply factors and patient perceptions.

Study goal:

Identify and analyze demand factors, supply factors and perceptions affecting BC patients' treatment choices, and model the demand function of BC patients in 5 key decision points: participation role in the decision making process, hospital choice, treatment regimen choice, surgical extent and surgeon choice.

Study hypothesis: Patient perceptions will have at least as much impact as demand and supply factors.

Study design:

Two stage study. A preliminary qualitative study, holding depth interviews with 20 breast cancer patients, 2 spouses and 3 staff members is taking place these days. The qualitative study findings will be used to develop a survey questionnaire for a cross sectional quantitative study, interviewing a quota sample of 425 breast cancer survivors, diagnosed up to 5 years prior to joining the study, who have successfully completed all radiation therapy and chemotherapy.

Data analysis:

Qualitative data will be analyzed according to the Criteria Bases Qualitative Methodology. Quantitative data will be analyzed by two-variable statistical analysis and multi-variable statistical analysis adjusted to the nature of the dependent and independent variables.

Possible policy recommendations:

Forming consulting teams for cancer patients. Improving medical information communication. Focusing patients on the key decisions they face. Evaluating patient needs using demand factors, supply factors and perceptions to create systemic tools helping them face treatment decisions.

ELIGIBILITY:
Inclusion Criteria:

* Hebrew speaking Jewish women
* Aged 30 - 75 years
* Diagnosed with breast cancer up to 5 years prior to study recruitment
* Successfully completed all chemotherapy and radiotherapy treatments
* Considered Cancer free

Exclusion Criteria:

* Any type of residual cancer
* Any type of chemotherapy or radiotherapy

Ages: 30 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hebrew speaking Jewish women aged 30 - 75 years, diagnosed with breast cancer up to 5 years prior to study recruitment, which have successfully completed all chemotherapy and radiotherapy treatments and are considered disease free.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2016-02; Primary Completion 2017-02 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Proportion of active, collaborative and passive patients according to the Control Preferences Scale | Through study completion, an average of 18 months.
  According to the Control Preferences Scale, a questionnaire developed by Degner and Colleagues (Degner, 1997), patients can take fully active role in the treatment decision process or be mostly active, collaborative, mostly passive or fully passive. The study will look at the factors and perceptions affecting patient's decision role.
Large or small hospital choice | Through study completion, an average of 18 months.
  The study interviews patients treated at two large Hospitals (Rambam, Sheba), and two small hospitals (Kaplan, Barzilay) looking for the factors and perceptions affecting large or small hospital choice.
Proportion of patients who chose an oncological regimen more intense than recommended by clinical guidelines. | Through study completion, an average of 18 months.
  The study will look at the factors and perceptions affecting patient's choice to undergo an oncological treatment more intense than recommended by clinical guidelines.
Proportion of patients choosing radical mastectomy over lumpectomy | Through study completion, an average of 18 months.
  The study will look at the factors and perceptions affecting patient's choice to undergo a surgical cancer removal procedure more radical than recommended by clinical guidelines.
Specific surgeon choice | Through study completion, an average of 18 months.
  The study will look at the factors and perceptions affecting patient's choice a specific surgeon in the Israeli healthcare system.

CONTACTS AND LOCATIONS:
Overall Officials: Shuli Brammli-Greenberg, PhD, Study Chair — Head of the Master of Public Health Program at Haifa University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Adams EK, Houchens R, Wright GE, Robbins J. Predicting hospital choice for rural Medicare beneficiaries: the role of severity of illness. Health Serv Res. 1991 Dec;26(5):583-612. PMID 1743970
- [Result] Beaver K, Luker KA, Owens RG, Leinster SJ, Degner LF, Sloan JA. Treatment decision making in women newly diagnosed with breast cancer. Cancer Nurs. 1996 Feb;19(1):8-19. doi: 10.1097/00002820-199602000-00002. PMID 8904382
- [Result] Benbassat J, Pilpel D, Tidhar M. Patients' preferences for participation in clinical decision making: a review of published surveys. Behav Med. 1998 Summer;24(2):81-8. doi: 10.1080/08964289809596384. PMID 9695899
- [Result] Bouche G, Migeot V, Mathoulin-Pelissier S, Salamon R, Ingrand P. Breast cancer surgery: do all patients want to go to high-volume hospitals? Surgery. 2008 Jun;143(6):699-705. doi: 10.1016/j.surg.2008.03.013. Epub 2008 May 9. PMID 18549885
- [Result] Celaya MO, Rees JR, Gibson JJ, Riddle BL, Greenberg ER. Travel distance and season of diagnosis affect treatment choices for women with early-stage breast cancer in a predominantly rural population (United States). Cancer Causes Control. 2006 Aug;17(6):851-6. doi: 10.1007/s10552-006-0025-7. PMID 16783613
- [Result] Duric V, Stockler M. Patients' preferences for adjuvant chemotherapy in early breast cancer: a review of what makes it worthwhile. Lancet Oncol. 2001 Nov;2(11):691-7. doi: 10.1016/S1470-2045(01)00559-9. PMID 11902540
- [Result] Harris KM. How do patients choose physicians? Evidence from a national survey of enrollees in employment-related health plans. Health Serv Res. 2003 Apr;38(2):711-32. doi: 10.1111/1475-6773.00141. PMID 12785569
- [Result] Hawley ST, Griggs JJ, Hamilton AS, Graff JJ, Janz NK, Morrow M, Jagsi R, Salem B, Katz SJ. Decision involvement and receipt of mastectomy among racially and ethnically diverse breast cancer patients. J Natl Cancer Inst. 2009 Oct 7;101(19):1337-47. doi: 10.1093/jnci/djp271. Epub 2009 Aug 31. PMID 19720966
- [Result] Jansen SJ, Otten W, Stiggelbout AM. Review of determinants of patients' preferences for adjuvant therapy in cancer. J Clin Oncol. 2004 Aug 1;22(15):3181-90. doi: 10.1200/JCO.2004.06.109. PMID 15284271
- [Result] Katz SJ, Lantz PM, Janz NK, Fagerlin A, Schwartz K, Liu L, Deapen D, Salem B, Lakhani I, Morrow M. Patient involvement in surgery treatment decisions for breast cancer. J Clin Oncol. 2005 Aug 20;23(24):5526-33. doi: 10.1200/JCO.2005.06.217. PMID 16110013
- [Result] Keating NL, Guadagnoli E, Landrum MB, Borbas C, Weeks JC. Treatment decision making in early-stage breast cancer: should surgeons match patients' desired level of involvement? J Clin Oncol. 2002 Mar 15;20(6):1473-9. doi: 10.1200/JCO.2002.20.6.1473. PMID 11896094
- [Result] Nelson JA, Tchou J, Domchek S, Sonnad SS, Serletti JM, Wu LC. Breast reconstruction in bilateral prophylactic mastectomy patients: factors that influence decision making. J Plast Reconstr Aesthet Surg. 2012 Nov;65(11):1481-9. doi: 10.1016/j.bjps.2012.05.001. Epub 2012 May 27. PMID 22640643
- [Result] Rees CE, Bath PA. The information needs and source preferences of women with breast cancer and their family members: a review of the literature published between 1988 and 1998. J Adv Nurs. 2000 Apr;31(4):833-41. doi: 10.1046/j.1365-2648.2000.01341.x. PMID 10759979
- [Result] Simes RJ, Coates AS. Patient preferences for adjuvant chemotherapy of early breast cancer: how much benefit is needed? J Natl Cancer Inst Monogr. 2001;(30):146-52. doi: 10.1093/oxfordjournals.jncimonographs.a003453. PMID 11773309
- [Result] Tropman SE, Ricketts TC, Paskett E, Hatzell TA, Cooper MR, Aldrich T. Rural breast cancer treatment: evidence from the Reaching Communities for Cancer Care (REACH) project. Breast Cancer Res Treat. 1999 Jul;56(1):59-66. doi: 10.1023/a:1006279117650. PMID 10517343
- [Result] Degner LF, Sloan JA, Venkatesh P. The Control Preferences Scale. Can J Nurs Res. 1997 Fall;29(3):21-43. PMID 9505581